CLINICAL TRIAL: NCT07071389
Title: Specific Supplementation in Counteracting the Adverse Effects of Oral Contraceptives
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The investigators were not able to recruit elegible patients and decided to halt the trial.
Sponsor: Lo.Li.Pharma s.r.l (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 000152
Record Dates: First submitted 2019-04-03; First posted 2025-07-17 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2019-04

CONDITIONS: Contraception
MeSH Terms: interventions — Contraceptives, Oral

STUDY DESIGN:
Intervention Model Description: Control group: oral contraceptive Study group: oral contraceptive + specific supplement
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (Active Comparator): Patients prescribed estroprogestinic oral contraceptive
  Interventions: Drug: Oral contraceptive
- Study group (Experimental): Patients prescribed estroprogestinic oral contraceptive were treatedwith Zyxelle supplement
  Interventions: Dietary Supplement: Zyxelle; Drug: Oral contraceptive

INTERVENTIONS:
Dietary Supplement: Zyxelle — Patients in the study group receive Zyxelle dietary supplement along with the oral contraceptive
  Arms: Study group
Drug: Oral contraceptive — Patients in the study group receive daily dose of estroprogestinic oral contraceptive

SUMMARY:
Prospective, controlled study. Administration of a specifically formulated supplement to women prescribed oral contraceptives. Evaluation of: a) reduction of adverse effects of the treatment; b) improvement of patients' quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Body Mass Index: 18-30 Kg/m2;
2. Prescription for COC treatment

Exclusion Criteria:

1. diabetes;
2. previous or existing breast pathologies;
3. hypertension;
4. obesity;
5. smoking habits;
6. cardiovascular disorders

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2018-01-08 (Actual); Primary Completion 2018-12-21 (Actual); Study Completion 2018-12-21 (Actual)

PRIMARY OUTCOMES:
cellulite | Change from baseline cellulite status at 3 months
  patients' self-assessed evaluation through a questionnaire
water retention | Change from baseline extracellular body water content at 3 months
  Bioelectrical impedance analysis (BIA)

SECONDARY OUTCOMES:
mood | Change from baseline mood at 3 months
  patients' self-assessed evaluation through a questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Studio Medico Anteo, Terni, TR, Italy

IPD SHARING:
Plan to Share IPD: No